CLINICAL TRIAL: NCT00275080
Title: A Phase 1 Study of Vorinostat (Suberoylanilide Hydroxamic Acid; SAHA) in Combination With Decitabine in Patients With Advanced Solid Tumors, Relapsed or Refractory Non-Hodgkin's Lymphoma, Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, or Chronic Myelogenous Leukemia in Blast Crisis
Brief Title: Vorinostat and Decitabine in Treating Patients With Advanced Solid Tumors or Relapsed or Refractory Non-Hodgkin's Lymphoma, Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00092; NCI-2009-00092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PMH-PHL-046; CDR0000456473; NCI-6869; PHL-046 (Other: Princess Margaret Hospital Phase 2 Consortium); 6869 (Other: CTEP); U01CA132123 (NIH)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-06

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Secondary Acute Myeloid Leukemia; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Blast Crisis; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Vorinostat; Decitabine

ARMS (1):
- Treatment (enzyme inhibitor, chemotherapy) (Experimental): Regimen 1 (sequential dosing): Patients receive oral vorinostat two or three times daily on days 6-21 or days 6-12 (patients with solid tumors or NHL only) and decitabine IV over 1 hour on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Regimen 2 (concurrent dosing): Patients receive oral vorinostat two or three times daily on days 1-21, days 1-14 (patients with hematological malignancies only), or two times daily on days 1-12 (patients with solid tumors or NHL only) and decitabine IV over 1 hour on days 1-5.
  Interventions: Drug: vorinostat; Drug: decitabine

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with decitabine in treating patients with advanced solid tumors or relapsed or refractory non-Hodgkin's lymphoma, acute myeloid leukemia, acute lymphocytic leukemia, or chronic myelogenous leukemia.

Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with decitabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the maximum tolerated dose and recommended phase II dose of vorinostat in conjunction with decitabine in patients with advanced solid tumors or relapsed or refractory non-Hodgkin's lymphoma, acute myeloid leukemia, acute lymphocytic leukemia, or chronic myelogenous leukemia in blast crisis.

SECONDARY OBJECTIVES:

I. Identify the minimal effective dose of vorinostat in conjunction with decitabine that will lead to DNA demethylation, histone acetylation, and gene reactivation with tolerable toxicity in these patients.

II. Determine the pharmacokinetic profiles of vorinostat and decitabine in these patients. Correlate pharmacokinetic profiles of vorinostat and decitabine with toxicity and biological activity in these patients.

III. Assess the antitumor activity of vorinostat and decitabine in these patients.

OUTLINE: This is a parallel group, multicenter, dose-escalation study of vorinostat. Patients are stratified according to disease (solid tumors or non-Hodgkin's lymphoma [NHL] vs hematological malignancies).

Patients receive 1 of 2 dosing regimens.

Regimen 1 (sequential dosing): Patients receive oral vorinostat two or three times daily on days 6-21 or days 6-12 (patients with solid tumors or NHL only) and decitabine IV over 1 hour on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Regimen 2 (concurrent dosing): Patients receive oral vorinostat two or three times daily on days 1-21, days 1-14 (patients with hematological malignancies only), or two times daily on days 1-12 (patients with solid tumors or NHL only) and decitabine IV over 1 hour on days 1-5.

Courses repeat every 28 days or 21 days (patients with hematological malignancies only) in the absence of disease progression or unacceptable toxicity. In both groups, cohorts of 3-6 patients receive escalating doses of vorinostat until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The dose level just below MTD would be declared the recommended phase II dose (RPTD). Up to 10 patients are treated at the RPTD. After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Confirmed relapsed or refractory acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) or chronic myelogenous leukemia in blast crisis (CML-BC)

    * Patients with acute promyelocytic leukemia who have relapsed while on tretinoin allowed
    * Patients with previously untreated AML who refuse induction chemotherapy allowed
    * Patients who are not candidates for aggressive management (those that have medical conditions that prevent the administration of standard curative chemotherapy or those who require an allogeneic bone marrow transplantation for curative therapy but lack an appropriate donor) are allowed
  * Histologically or cytologically confirmed relapsed or refractory non-Hodgkin's lymphoma (NHL)
  * Histologically confirmed solid tumor that is metastatic or unresectable or for which standard curative or palliative measures do not exist or are no longer effective

    * Clinically or radiologically documented disease
    * Patients whose only evidence of disease is tumor marker elevation are not eligible
* Patients with AML, ALL, or CML-BC who have cerebral spinal fluid involvement may be included

  * May be treated with intrathecal cytarabine and/or methotrexate prior to and/or during the study
* No known brain metastases in patients with solid tumors or NHL
* ECOG performance status 0-2
* Karnofsky 60-100%
* Life expectancy > 12 weeks for patients with solid tumors (including non-Hodgkin's lymphoma) and 6 weeks for patients with hematological malignancies
* Patients with solid tumors (including NHL) must also have normal marrow function as defined below:

  * Leukocytes ≥ 3,000/mm^3
  * Absolute neutrophil count ≥ 1,500/mm^3
  * Platelets ≥ 100,000/mm^3
* Creatinine ≤ 150 μmol/L
* Creatinine clearance ≥ 60 mL/min
* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control or abstinence) prior to study entry and for the duration of study participation
* Not pregnant or nursing
* Negative pregnancy test
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or other agents used in study
* Able to take oral medications
* Patients who have a clinical or radiological diagnosis of bowel obstruction are ineligible
* No ongoing or active infection
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No psychiatric illness/social situations that would limit compliance with study requirements
* No other uncontrolled intercurrent illness
* No limitation on the number or types of prior therapy
* At least 3 weeks since prior radiotherapy, chemotherapy (6 weeks for nitrosoureas or mitomycin C), or molecularly targeted agents

  * Exceptions may be made for low-dose, non-myelosuppressive radiotherapy
* At least 2 weeks since prior valproic acid or any other histone deacetylase inhibitor
* Must have recovered from prior therapy
* Patients with hematological malignancies may receive hydroxyurea until 24 hours prior to starting study medications
* Previous surgery is permitted provided that wound healing has occurred
* No prior decitabine
* No other concurrent investigational agents
* No other concurrent investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy
* No HIV-positive patients receiving combination antiretroviral therapy
* No concurrent prophylactic hematopoietic growth factors (e.g. filgrastim [G-CSF], sargramostim [GM-CSF], thrombopoietin, or epoetin alfa)

  * Hematopoietic growth factors colony stimulating factors for the treatment of cytopenia may be permitted at the discretion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-02; Primary Completion 2009-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose of vorinostat and decitabine | Course 1
  Graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

SECONDARY OUTCOMES:
Minimal effective dose of vorinostat in combination with decitabine by bone marrow and/or peripheral blood (for leukemia) | Baseline and between days 3-10
Pharmacokinetics of vorinostat in conjunction with decitabine | Days 1-15
  Measured by peripheral blood. Performed by high-performance liquid chromatography (HPLC). Estimated by taking the mean concentration one hour after administration per patient on days 1 and 5 and estimating the mean, median and range over all patients.
Antitumor activity | Every 4 weeks for leukemia and every 8 weeks for solid tumors or NHL
  Measured by Response Evaluation Criteria In Solid Tumors (RECIST), NCI-international working group (IWG), and NCI criteria.
Methylation status of gene promoter regions and gene expression | Baseline and between days 3-10
  Measured by bone marrow and/or peripheral blood.
Altered response of leukemic cells to PPAr and RAR ligands | Baseline and between days 3-8
  Collected by bone marrow and/or peripheral blood (for leukemia)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yee, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (4):
- Canada (4):
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario